CLINICAL TRIAL: NCT01027988
Title: Retina Microvascularisation and Cardiovascular Heart Disease Prediction
Status: Completed | Type: Observational
Sponsor: Montreal Heart Institute (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government)
Responsible Party: Principal Investigator, Bernard Thibault, Cardiologist - Electrophysiologist, Montreal Heart Institute
Other Study IDs: ICM 08-1050
Record Dates: First submitted 2009-12-07; First posted 2009-12-09 (Estimated); Last update posted 2013-10-30 (Estimated); Status verified 2013-10

CONDITIONS: Cardiovascular Disease
Keywords: Retinal Microvascularisation; Fundus; mfERGs; CHF; Cardiovascular Disease; Coronarography; Macrovascularisation; The objectives are to assess if if any retinal vascular disorder in arterioles and venules can be predictive for cardiovascular morbidity and mortality
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Earlier studies have found that retinal photography could be very useful for evaluating the condition of microcirculation and the risk of cardiovascular diseases in patients. The architectural changes in retinal vascularisation strongly correlates with macrovascular remodeling. Also, recent founding suggests a possible close anatomical parallel between both the macrovascular and the microvascular blood.

Our objectives are to assess (1) in which age and sex subgroups, if any, retinal vascular alteration in arterioles and venules can be predictive for cardiovascular morbidity and mortality; and (2) whether variations in arteriolar or venular caliber will predict better cardiovascular pathogenesis in normal and patient population. If the association between the diameter of the retinal vessels and the risks of cardiovascular disease is verified during this study, the impact on prevention would be enormous. The retinal microvascular change could become a powerful biomarker in the early detection of the cardiovascular pathogenesis and death risk

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 to 70 years old (male/female)
* indication of coronarography within the last 3 month preceding the enrollment
* Patients with history of stroke, heart failure or arteriosclerosis.
* At least one of the following risk factors for cardiovascular complication:

  * Hypertension
  * Coronary heart disease (CHD)
  * Diabetes
  * Structural heart disease
  * Dyslipidemia
  * Obesity

Exclusion Criteria:

* Patients with a permanent pacemaker or ICD
* Nephrosis or chronic renal failure
* The study interferes with therapeutic or diagnostic procedures
* Patients with inability to consent or comply with follow up requirements
* Patients with glaucoma
* Patients with any retina degeneration disease vascular age-related macular degeneration or any -retina degeneration disease
* Patients who are pregnant

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: (50 to 70 years old) with history of coronary heart disease (CHD) or one or more risk factors.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Occurrence of a major cardiovascular event or complication, defined as hospitalization, death from coronary heart disease, hypertension, arteriosclerosis, nonfatal non-procedure-related myocardial infarction, or fatal or nonfatal stroke | 2 years

SECONDARY OUTCOMES:
Characterization of any retinal vascular disorders occurring at any time during the study: i. Confirmed by an ophthalmologist examination and either an fundus camera or an mfERGs examination ii. Occurrence of serious ophthalmic event | 2 years
Correlation with possible cardiovascular event | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Thibault, MD, Principal Investigator — Montreal Heart Institute
Locations (1):
- Montreal Heart Institute, 5000 Belanger Street, Montreal, Quebec, Canada